CLINICAL TRIAL: NCT00620412
Title: Lactobacillus GG to Enhance the Immunogenicity of Influenza Vaccine in Healthy Adults - Proof of Concept Study
Brief Title: Probiotics to Enhance Immunogenicity of Influenza Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Amerifit Brands Inc (Industry)
Responsible Party: Patricia L. Hibberd, MD, PhD, Tufts Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 7142
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Healthy
Keywords: influenza; vaccines; probiotics; LGG
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment (Active Comparator)
  Interventions: Dietary Supplement: Lactobacillus rhamnosus; Biological: Influenza Virus Vaccine Live, Intranasal
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo control; Biological: Influenza Virus Vaccine Live, Intranasal

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus — 2 capsules by mouth 2 times a day for 28 days. Each capsule contains 1x10^10 LGG organisms.
  Other Names: Culturelle
  Arms: treatment
Dietary Supplement: placebo control — 2 capsules by mouth twice a day for 28 days
  Arms: placebo
Biological: Influenza Virus Vaccine Live, Intranasal — intranasal spray, 0.1ml per nostril, one time dose
  Other Names: FluMist

SUMMARY:
The purpose of this study is to determine whether the food supplement called Lactobacillus rhamnosus GG (LGG) may help boost the effectiveness of the nasal flu vaccine. Preliminary data from several studies of healthy volunteers suggest that LGG boosts the immune response to vaccines. Fifty-two subjects will be recruited into the study, all will receive the nasal flu vaccine. Twenty-six will receive capsules that contain LGG, 26 will receive placebo capsules. Blood and nasal specimens will be collected weekly for four weeks and at eight weeks to evaluate the initial mucosal and systemic immune response to the immunization. This study will provide preliminary data on whether the immune response of healthy adults to the nasal influenza vaccine can be boosted by LGG.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-49 years
* Available for clinic visits at Tufts-New England Medical Center
* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) obtained
* Ability of participant to understand and comply with the requirements of the protocol

Exclusion Criteria:

* History of any medical conditions for which the CDC states should not be vaccinated with LAIV (asthma, reactive airways disease, other chronic disorders of the pulmonary or cardiovascular systems; metabolic diseases such as diabetes, renal dysfunction, and hemoglobinopathies; or persons with known or suspected immunodeficiency diseases)
* Self-reported vaccination with the influenza vaccine for the current influenza season (2007-8); vaccination with any vaccine within the one month period prior to study enrollment or intent to receive any other vaccine during the study period; hypersensitivity to any influenza vaccine components including thimersol or egg or Guillain-Barre syndrome
* Self-reported treatment with immunomodulator/immunosuppressor drugs (interleukins, corticosteriods (oral or inhaled)), G(M)-CSF in 4 weeks before enrollment or self-reported history of IL-2 administration within 5 years; use of theophylline preparations or warfarin because of the theoretical possibilities of enhanced drug effects and toxicities following influenza vaccination; medication use that might affect the immune response to a vaccine or effects of LGG (no antibiotics during the previous 4 weeks)
* Current alcohol, substance abuse, or systemic/psychiatric illness that potentially could interfere with compliance and ability to make study visits
* Health care or day care workers or close contacts with immunosuppressed persons because of the theoretical risk that LAIV could be transmitted to the immunosuppressed person and cause disease, per CDC recommendations
* Use of LGG or other probiotics in 4 weeks before enrollment. Yogurt consumption is not an exclusion criteria, but subjects will be asked to avoid consumption of other lactobacilli and probiotic organisms during the study period
* Abnormalities upon physical examination
* Acute febrile illness on day of intended immunization - immunization deferred until illness resolved
* Routine laboratory tests outside the limits outlined for this study:

  1. hemoglobin >=11.5g/dL for women; >=13.5 g/dL for men
  2. WBC 3,300-12,000 cells/mm^3
  3. Differential within normal range
  4. Platelets 125,000-550,000 /mm^3
  5. ALT <= upper limit of normal
  6. Serum creatinine <= upper limit of normal
  7. Normal urinalysis (negative glucose, negative or trace protein, and negative or trace hemoglobin)
  8. Negative beta-HCG pregnancy test (urine or serum) for women presumed to be of reproductive potential because LAIV is contraindicated in pregnant women
  9. negative HIV test
  10. negative hepatitis B surface antigen
  11. negative anti-HCV

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To measure anti-influenza systemic and mucosal antibody responses 4 weeks after administration of influenza vaccine (LAIV) to healthy subjects aged 18-49 and to compare responses in subjects receiving Lactobacillus GG (LGG) versus placebo | 4 weeks

SECONDARY OUTCOMES:
To assess time course of antibody response after administration of influenza vaccine (LAIV) and to compare responses in subjects receiving LGG versus placebo | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L Hibberd, MD, PhD, Principal Investigator — Tufts Medical Center

REFERENCES:
- [Derived] Davidson LE, Fiorino AM, Snydman DR, Hibberd PL. Lactobacillus GG as an immune adjuvant for live-attenuated influenza vaccine in healthy adults: a randomized double-blind placebo-controlled trial. Eur J Clin Nutr. 2011 Apr;65(4):501-7. doi: 10.1038/ejcn.2010.289. Epub 2011 Feb 2. PMID 21285968